CLINICAL TRIAL: NCT03474263
Title: A Phase 2a, Open-Label Biomarker Study of IC14 for the Treatment of Patients With
Brief Title: IC14 for Rapidly Progressive Amyotrophic Lateral Sclerosis (ALS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: seeking research grant support
Sponsor: Implicit Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS02
Record Dates: First submitted 2018-03-09; First posted 2018-03-22 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Motor Neurone Disease (MND); Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Open-label Biomarkers-Driven Study Historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IC14 (monoclonal anti-CD14 antibody) (Experimental): Biologic: IC14 (monoclonal anti-CD14 antibody) 4 mg/kg intravenously followed by IC14 2 mg/kg intravenously on Days 2-4. This four-day cycle will be repeated on Days 8-11.
  Interventions: Biological: Biologic: IC14 (monoclonal antibody against human CD14)

INTERVENTIONS:
Biological: Biologic: IC14 (monoclonal antibody against human CD14) — IC14 intravenous infusion daily for four days on two successive weeks then MR-PET Scan evaluation for impact on glial activation.
  Other Names: Anti-CD14

SUMMARY:
Patients with rapidly progressive ALS will be assigned to IC14 intravenously on Day 1-4. This 4-day course will be repeated on Days 8-11. Patients will all undergo MR-PET scans at two time points: before treatment onset and after the last treatment cycle. This scan will measure areas of ALS disease activity and assess response to IC14 treatment. MR-PET scans will be compared to historical controls.

DETAILED DESCRIPTION:
This is an open-label, biomarkers-driven study.

Patients with rapidly progressive ALS will be assigned to the following dose regimen of IC14:

• 4 mg/kg intravenously on Day 1, followed by 2 mg/kg daily x 3 days on Days 2-4. This 4-day course will be repeated on Days 8-11.

Patients will be followed for 28 days after the last dose of study drug. Patients will all undergo [11C]-PBR28-MR-PET scans at two time points: before treatment onset and after the last treatment cycle.

Patients will be followed for 28 days after the last dose of study drug for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing informed consent and informed consent form signed prior to initiation of any study-specific procedures.
2. Familial or sporadic ALS defined as clinically possible, probable, or definite by El Escorial Criteria.
3. Rapidly progressive ALS defined by the Revised ALS Functional Rating Scale (ALSFRS-R) slope ≥1 (48 minus ALSFRS-R score at screening / disease duration in months ≥ 1).
4. Upper Motor Neuron Burden Score of ≥ 25 (out of 45) at screening
5. First symptoms of ALS within 3 years of the screening visit
6. Age between 18 and 80 years at the time of the screening visit.
7. Not taking riluzole or edaravone or on a stable dose of riluzole or edaravone for at least 3 months prior to screening visit.
8. Adequate bone marrow reserve, renal and liver function:

   1. absolute neutrophil count ≥ 1500/µL
   2. lymphocyte count < 6000/µL
   3. platelet count ≥ 150,000/µL
   4. hemoglobin ≥ 11 g/dL
   5. creatinine clearance ≥ 60 mL/min
   6. alanine transaminase (ALT) and/or aspartate transaminase (AST) ≤ 3x upper limits of normal (ULN)
   7. total bilirubin ≤ 1.5x ULN
   8. serum albumin ≥ 2.8 g/dL
9. Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods:

   1. Sexual abstinence (inactivity) for 1 month prior to screening through study completion; or
   2. Intrauterine device (IUD) in place for at least 3 months prior to study through study completion; or
   3. Stable hormonal contraception for at least 3 months prior to study through study completion; or
   4. Surgical sterilization (vasectomy) of male partner at least 6 months prior to study.
10. To be considered of non-childbearing potential, females should be surgically sterilized (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be post-menopausal and at least 3 years since last menses.
11. Males with female partners of childbearing potential must use contraception through study completion.
12. Ability to safely lie flat for 90 min for magnetic resonance-positron emission tomography (MR-PET) procedures in the opinion of the Investigator.
13. Patients must also have a genotype associated with a high or mixed affinity translocator protein (TSPO) (Ala/Ala or Ala/Thr) and ability to safely undergo MR-PET scans based on the opinion of the Investigator.

Exclusion Criteria:

1. Dependence on invasive or non-invasive ventilation, defined as being unable to lay supine without it, unable to sleep without it, or continuous daytime use; presence of tracheostomy at screening; or presence of diaphragm pacing system at screening.
2. Exposure to any experimental treatment for ALS within the last 30 days or five half-lives, whichever is longer.
3. Treatment within 12 months with immunomodulator or immunosuppressant agent (including but not limited to cyclophosphamide, cyclosporine, interferon-α, interferon-β-1a, rituximab, alemtuzumab, azathioprine, etanercept, infliximab, adalimumab, certolizumab, golimumab, anakinra, rilonacept, secukinumab, tocilizumab, mycophenolate mofetil, methotrexate, cell-depleting agents, total lymphoid irradiation, dimethyl fumarate). Treatment with intravenous immunoglobulin (IVIG) within 2 months. Non-steroidal anti-inflammatory drugs (NSAIDs) are acceptable.
4. Exposure at any time to any cell or gene therapies under investigation for the treatment of ALS.
5. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other opportunistic infections; or major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 4 weeks.
6. Live-attenuated vaccines within 30 days before dosing. Subjects must agree to forego live-attenuated vaccines throughout the study, including 60 days after the last dose of study drug.
7. History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
8. History of one or more of the following: cardiac insufficiency (New York Heart Association [NYHA] III/IV), uncontrolled cardiac arrhythmias, unstable ischemic heart disease, or uncontrolled hypertension (systolic blood pressure > 170 mmHg or diastolic blood pressure > 110 mmHg).
9. History of myocardial infarction, or cerebrovascular accident.
10. Unstable pulmonary, renal, hepatic, endocrine or hematologic disease.
11. Autoimmune disease, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis.
12. Evidence of active malignant disease, malignancies diagnosed within the previous 5 years, or breast cancer diagnosed within the previous 5 years (except skin cancers other than melanoma).
13. History of human immunodeficiency virus infection or other immunodeficiency illness.
14. Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days.
15. History of drug abuse (not including marijuana use) or alcoholism within the past 12 months.
16. Significant neuromuscular disease other than ALS.
17. Other ongoing disease that may cause neuropathy, such as toxin exposure, dietary deficiency, uncontrolled diabetes, hyperthyroidism, cancer, systemic lupus erythematosus or other connective diseases, infection with HIV, hepatitis B virus (HBV), or hepatitis C (HCV), Lyme disease, multiple myeloma, Waldenström's macroglobulinemia, amyloid, and hereditary neuropathy.
18. Pregnancy or breastfeeding.
19. Deprivation of freedom by administrative or court order.
20. Any contraindication to undergo magnetic resonance imaging (MRI) studies such as history of a cardiac pacemaker or pacemaker wires; metallic particles in the body; vascular clips in the head; prosthetic heart valves; or severe claustrophobia.
21. Unwilling or unable to discontinue benzodiazepine usage [other than lorazepam (Ativan®), clonazepam (Klonopin®), or zolpidem (Ambien®)] for one day prior to and during scanning.
22. Research imaging-related radiation exposure exceeds current institutional Radiology Department guidelines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-04-12 (Estimated); Study Completion 2021-07-12 (Estimated)

PRIMARY OUTCOMES:
Glial Activation | one month
  Glial activation measured in the motor region measured by [11C]-PBR28 positron emission tomography (PET). Studies have shown this marker localizes to areas of glial activation and correlates with disease progression and outcomes.
Serum neurofilament | one month
  Serum neurofilament is a biomarker that has been shown to correlate with ALS severity
Urinary p75 neurotrophin receptor | one month
  Urinary p75 neurotrophin receptor is a biomarker that has been shown to correlate with ALS severity

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety, Tolerability) | six weeks
  Adverse event reporting
Immunogenicity | six weeks
  Human anti-monoclonal antibodies
Peak Plasma Concentration of IC14 | one month
  Peak Plasma Concentration (Cmax) of IC14
Pharmacodynamics | one month
  Monocyte CD14 saturation

CONTACTS AND LOCATIONS:
Overall Officials: Jan Agosti, MD, Principal Investigator — Implicit Bioscience Ltd.
Locations (1):
- Royal Brisbane & Women's Hospital, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No